CLINICAL TRIAL: NCT01737502
Title: A Phase I-II Trial of Combined PKCι and mTOR Inhibition for Patients With Advanced or Recurrent Lung Cancer (NSCLC and SCLC) Without Standard Treatment Options
Brief Title: Sirolimus and Auranofin in Treating Patients With Advanced or Recurrent Non-Small Cell Lung Cancer or Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1125; NCI-2012-00518 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 11-001987 (Other: Mayo Clinic Institutional Review Board); R21CA153000 (NIH)
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Results first posted 2025-08-20 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2024-03

CONDITIONS: Extensive Stage Small Cell Lung Carcinoma; Lung Adenocarcinoma; Recurrent Non-Small Cell Lung Carcinoma; Recurrent Small Cell Lung Carcinoma; Squamous Cell Lung Carcinoma; Stage IIIA Non-Small Cell Lung Cancer; Stage IIIB Non-Small Cell Lung Cancer; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Auranofin; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (auranofin and sirolimus) (Experimental): Patients receive auranofin PO on days 1-28 and sirolimus PO on days 1-28 (days 8-28 of course 1). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Auranofin; Drug: Sirolimus; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Auranofin — Given PO
  Other Names: Ridaura
Drug: Sirolimus — Given PO
  Other Names: AY 22989; RAPA; SILA 9268A; WY-090217
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of auranofin when given together with sirolimus and to see how well it works in treating patients with lung cancer that has spread or other places in the body and cannot be cured or controlled by treatment or has come back after a period of time during which the cancer could not be detected. Auranofin and sirolimus may stop or slow the growth of lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the maximum tolerated dose of auranofin plus sirolimus after at least one line of platinum based chemotherapy for lung cancer (squamous, ras-mutated adenocarcinoma, or small cell lung cancer) patients with no acceptable standard treatment options. (Phase I) II. To assess the progression-free survival at four months of patients treated with auranofin after at least one line of platinum based chemotherapy for lung cancer (squamous, ras-mutated adenocarcinoma, or small cell lung cancer) patients with no acceptable standard treatment options. (Phase II)

SECONDARY OBJECTIVES:

I. To assess the overall survival in this population in comparison to recent historical controls.

II. To determine the adverse events (AE) profile and safety of the regimen. III. To determine the overall response rate, per Response Evaluation Criteria In Solid Tumors (RECIST) criteria, and duration of tumor response in those patients with measurable disease.

TERTIARY OBJECTIVES:

I. To assess the relationship between molecular correlates and progression-free survival (PFS), overall survival (OS), response and adverse events.

OUTLINE: This is a phase I, dose-escalation study of auranofin followed by a phase II study.

Patients receive auranofin orally (PO) on days 1-28 and sirolimus PO on days 1-28 (days 8-28 of course 1). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3-6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic confirmation of lung cancer (squamous, ras-mutated adenocarcinoma or small cell lung cancer)
* Patients must have received at least one course of chemotherapy consisting of a platinum doublet and must have no acceptable standard treatment options
* Prior radiation therapy is permitted as long as:

  * Recovered from the toxic effects of radiation treatment before study entry, except for alopecia
* Absolute neutrophil count (ANC) >= 1500 uL
* Platelets (PLT) >= 100,000 uL
* Hemoglobin (Hgb) >= 9 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN) or direct bilirubin =< ULN
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamic pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) =< 3 x ULN or SGOT (AST) and SGPT (ALT) =< 5 x ULN is acceptable if liver has tumor involvement
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, 2
* Negative serum pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Ability to provide informed consent
* Life expectancy >= 12 weeks
* Willing to return to Mayo Clinic enrolling institution for follow-up
* Willing to provide tissue samples for correlative research purposes

Exclusion Criteria:

* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Symptomatic, untreated, or uncontrolled central nervous system (CNS) metastases or seizure disorder; NOTE: patients with treated CNS metastases without evidence of progression and without uncontrolled symptoms or need for steroids may enroll
* Human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy are excluded
* Unwilling or unable to, comply with the protocol
* Any of the following prior therapies:

  * Radiation to >= 25% of bone marrow
  * Major surgery (i.e., laparotomy), open biopsy, or significant traumatic injury =< 4 weeks prior to registration; minor surgery =< 2 weeks prior to registration; insertion of a vascular access device is not considered major or minor surgery in this regard
* Any of the following concurrent severe and/or uncontrolled medical conditions:

  * Hypertension, labile hypertension, or history of poor compliance with antihypertensive medication
  * Angina pectoris
  * History of congestive heart failure =< 3 months, unless ejection fraction > 40%
  * Myocardial infarction =< 6 months prior to registration
  * Cardiac arrhythmia
  * Poorly controlled diabetes
  * Interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
  * Active or recent history of hemoptysis; if hemoptysis has resolved with measures such as palliative radiation therapy (e.g. 3000 cGy over 10 fractions), arteriographic embolization or endobronchial interventions (e.g. photodynamic therapy, brachytherapy), etc. for > 14 days, patients may be considered for participation in this study
  * >= Grade 2 hypertriglyceridemia
  * >= Grade 2 hypercholesterolemia
  * Any illness that in the opinion of the investigator would compromise the ability of the patient to participate safely in the clinical trial
* Use of St. John's Wort because of its effects on hepatic drug metabolism
* Other active malignancy: EXCEPTIONS: Non-melanoma skin cancer, localized prostate cancer, or carcinoma-in-situ of the cervix; NOTE: If there is a history or prior malignancy, patient must not be receiving other cytotoxic or molecularly targeted therapeutics treatment for their cancer; patients receiving certain hormonal manipulations as part of their treatment may be allowed to continue at the discretion of the Principal Investigator (PI) (e.g. luteinizing hormone-releasing hormone [LHRH] analogs for prostate cancer)
* Unable to discontinue use of potent cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inhibitors/inducers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-05-14 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yanyan Lou, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida

REFERENCES:
- [Derived] Jatoi A, Foster NR, Wahner Hendrickson A, Block MS, Weroha SJ, Asmus EJ, Murray NR, Fields AP. A Phase 2 Trial of Protein Kinase C Iota Inhibition With the Combination of Auranofin and Sirolimus in Patients With Recurrent Ovarian Cancer. Am J Clin Oncol. 2025 Oct 20. doi: 10.1097/COC.0000000000001263. Online ahead of print. PMID 41114938
- [Derived] Rousselle B, Massot A, Privat M, Dondaine L, Trommenschlager A, Bouyer F, Bayardon J, Ghiringhelli F, Bettaieb A, Goze C, Paul C, Malacea-Kabbara R, Bodio E. Conception and Evaluation of Fluorescent Phosphine-Gold Complexes: From Synthesis to in vivo Investigations. ChemMedChem. 2022 Jun 3;17(11):e202100773. doi: 10.1002/cmdc.202100773. Epub 2022 Mar 29. PMID 35254001
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 0: Patients receive 3mg auranofin PO on days 1-28 and sirolimus PO on days 1-28 (days 8-28 of course 1). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  >
  > Auranofin: Given PO
  >
  > Sirolimus: Given PO
  >
  > Laboratory Biomarker Analysis: Correlative studies
  >
  > Pharmacological Study: Correlative studies
- Dose Level 1: Patients receive 6mg auranofin PO on days 1-28 and sirolimus PO on days 1-28 (days 8-28 of course 1). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  >
  > Auranofin: Given PO
  >
  > Sirolimus: Given PO
  >
  > Laboratory Biomarker Analysis: Correlative studies
  >
  > Pharmacological Study: Correlative studies
Period: Phase I
Arm/Group | Dose Level 0 | Dose Level 1
Started | 3 | 3
Completed | 0 | 0
Not Completed | 3 | 3
Not completed — Disease progression | 2 | 3
Not completed — Complicating disease | 1 | 0
Period: Phase II
Arm/Group | Dose Level 0 | Dose Level 1
Started | 0 | 23
Completed | 0 | 0
Not Completed | 0 | 23
Not completed — Adverse Event | 0 | 3
Not completed — Disease progression | 0 | 18
Not completed — Death | 0 | 1
Not completed — Transition to hospice care | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 0: Patients receive 3mg auranofin PO on days 1-28 and sirolimus PO on days 1-28 (days 8-28 of course 1). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. > > Auranofin: Given PO > Sirolimus: Given PO > Laboratory Biomarker Analysis: Correlative studies > Pharmacological Study: Correlative studies
- Dose Level 1: Patients receive 6mg auranofin PO on days 1-28 and sirolimus PO on days 1-28 (days 8-28 of course 1). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. > > Auranofin: Given PO > Sirolimus: Given PO > Laboratory Biomarker Analysis: Correlative studies > Pharmacological Study: Correlative studies
- Total: Total of all reporting groups
Arm/Group | Dose Level 0 | Dose Level 1 | Total
Number analyzed (Participants) | 3 | 26 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (7.8) | 62.38 (9.3) | 61.52 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 12 | 14
  Male | 1 | 14 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 24 | 27
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 24 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 26 | 29
Histologic Type [Count of Participants; unit: Participants]
  Small cell lung cancer | 0 | 9 | 9
  Non-small cell lung cancer | 2 | 17 | 19
  Unknown | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Phase 1 Patients Experiencing a DLT
Description: The number and severity of all adverse events (overall and by dose level) will be tabulated and summarized. A DLT is defined as an adverse event during the first cycle of, at least possibly related to study treatment, and one of the following: Grade 4 Neutropenia, Grade 4 Thrombocytopenia, ≥Grade 3 Anaphylaxis, ≥Grade 3 Proteinuria, ≥Grade 3 Hematuria, ≥Grade 3 Rash acneiform, ≥Grade 3 Diarrhea, ≥Grade 3 Mucositis oral
Time Frame: 28 days
Population: Only phase 1 patients were included in analysis
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 0: Patients receive 3mg auranofin PO on days 1-28 and sirolimus PO on days 1-28 (days 8-28 of course 1). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. > > Auranofin: Given PO >
  * Sirolimus: Given PO >
  * Laboratory Biomarker Analysis: Correlative studies >
  * Pharmacological Study: Correlative studies
- Dose Level 1: Patients receive 6mg auranofin PO on days 1-28 and sirolimus PO on days 1-28 (days 8-28 of course 1). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. > > Auranofin: Given PO >
  * Sirolimus: Given PO >
  * Laboratory Biomarker Analysis: Correlative studies >
  * Pharmacological Study: Correlative studies
Arm/Group | Dose Level 0 | Dose Level 1
Number analyzed (Participants) | 3 | 3
Participants | 0 | 0

2. Primary Outcome: Number Phase 1 Patients Experiencing a Grade 3+ AE
Description: Number and severity of all adverse events (overall and by dose level) will be tabulated and summarized.
Time Frame: Up to 5 years
Population: Only phase 1 patients were included in analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 0 | Dose Level 1
Number analyzed (Participants) | 3 | 3
Participants | 2 | 1

3. Primary Outcome: Progression-free Survival Rate
Description: A patient is considered to be a 4-month progression-free survivor, or success, if the patient is 4 months from registration without a documentation of disease progression. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Confidence intervals for the true success proportion will be calculated using the properties of the binomial distribution. Additionally, an estimate and confidence interval for the 4-month progression-free survival rate incorporating censoring may be computed using the method of Kaplan-Meier.
Time Frame: 4 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Level 0 | Dose Level 1
Number analyzed (Participants) | 3 | 26
percentage of participants | 66.7 [9.4 to 99.2] | 28.0 [12.1 to 49.4]

4. Secondary Outcome: Overall Survival Time
Description: Overall Survival (OS) is defined as the length of time from study enrollment until death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Level 0 | Dose Level 1
Number analyzed (Participants) | 3 | 26
months | 4.9 [3.6 to NA] — Upper limit of the 95% Confidence Interval was not estimable due to an insufficient number of participants with events. | 8.6 [7.5 to 11.7]

5. Secondary Outcome: Progression-free Survival Time
Description: Progression-free survival is defined as the time from study enrollment until disease progression or death from any cause. The distribution of progression-free survival time will be estimated using the method of Kaplan-Meier.
Time Frame: up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Level 0 | Dose Level 1
Number analyzed (Participants) | 3 | 26
months | 4.9 [1.7 to NA] — Upper limit of the 95% Confidence Interval was not estimable due to an insufficient number of participants with events | 2.1 [1.8 to 4.2]

6. Secondary Outcome: Number of Patients Achieving a Complete Response (CR) or Partial Response (PR) Noted as the Objective Status
Description: The overall response rate will be estimated in the subset of patients with measurable disease by the number of responses in evaluable patients with measurable disease divided by the total number of evaluable patients with measurable disease.
Time Frame: Up to 5 years
Population: Only patients with measurable disease were included in analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 0 | Dose Level 1
Number analyzed (Participants) | 3 | 21
Participants | 1 | 2

7. Secondary Outcome: Duration of Response
Description: Defined for all evaluable patients with measurable disease who have achieved a response as the date at which the patient's earliest best objective status is first noted to be a CR or PR to the earliest date progression is documented. The distribution of duration of response will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 5 years
Population: Only patients that achieved a CR or PR for a known amount of time were included in analysis
Measure: Mean (Full Range); unit: months
Arm/Group | Dose Level 0 | Dose Level 1
Number analyzed (Participants) | 0 | 2
months |  | 16.25 [14.7 to 17.8]

8. Other Pre Specified Outcome: Change in Protein Kinase C (PKC) Iota Protein Expression
Description: Will be evaluated at baseline using the baseline tissue specimen and explored in relation to 4-month progression-free survival and subsequently in relation to other clinical outcomes such as tumor response and adverse event incidence using two-way tables and analyzed using Fisher's exact tests.
Time Frame: Baseline to up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 5 years
Groups:
- Dose Level 0: Patients receive 3mg auranofin PO on days 1-28 and sirolimus PO on days 1-28 (days 8-28 of course 1). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  * Auranofin: Given PO
  * Sirolimus: Given PO
  * Laboratory Biomarker Analysis: Correlative studies
  * Pharmacological Study: Correlative studies
- Dose Level 1: Patients receive 6mg auranofin PO on days 1-28 and sirolimus PO on days 1-28 (days 8-28 of course 1). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  * Auranofin: Given PO
  * Sirolimus: Given PO
  * Laboratory Biomarker Analysis: Correlative studies
  * Pharmacological Study: Correlative studies
Arm/Group | Dose Level 0 | Dose Level 1
All-Cause Mortality (participants affected / at risk) | 1/3 | 3/26
Serious Adverse Events (participants affected / at risk) | 2/3 | 8/26
Other Adverse Events (participants affected / at risk) | 3/3 | 23/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 0 (N=3) | Dose Level 1 (N=26)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Death NOS (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 0 (0) | 2 (2)
Lung infection (Infections and infestations) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 0 (N=3) | Dose Level 1 (N=26)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 18 (85)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 17 (47)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 2 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 12 (17)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3)
Edema limbs (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 2 (3)
Fever (General disorders) | 0 (0) | 3 (3)
Bladder infection (Infections and infestations) | 0 (0) | 1 (2)
Bronchial infection (Infections and infestations) | 1 (1) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (2) | 0 (0)
Papulopustular rash (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (2)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0)
Cholesterol high (Investigations) | 1 (1) | 13 (41)
Creatinine increased (Investigations) | 1 (1) | 3 (21)
Platelet count decreased (Investigations) | 2 (2) | 5 (10)
Weight loss (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 7 (14)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2) | 13 (53)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (15)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (20)
Dizziness (Nervous system disorders) | 1 (1) | 4 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 5 (14)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/02/NCT01737502/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-28): https://cdn.clinicaltrials.gov/large-docs/02/NCT01737502/ICF_001.pdf